CLINICAL TRIAL: NCT03625271
Title: A Prospective Study to Evaluate the Utility, Safety, and Efficacy of Using PEER Interactive to Inform the Prescription of Medications to Subjects With a Primary Diagnosis of a Depressive Disorder and Comorbidity of Non-psychotic Behavioral Disorders
Brief Title: The Canadian Armed Forces PEER Study
Acronym: PEERCanada
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MYnd Analytics (Industry)
Collaborators: University of Ottawa (Other); Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS013
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Depression; Non-psychotic Diagnosis as Co-morbidity
Keywords: Electroencephalogram; data base; machine learning
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Blinded participants will be randomized into a control or experimental group and receive a quantitative electroencephalogram (QEEG). Experimental group clinicians will use the PEER Interactive Report in the medication prescription process. Control group clinicians will not receive an Outcome Report. For the experimental group the clinician is expected to incorporate the guidance of the subject's PEER Outcome Report. Study staff will note the basis for all medication decisions in the subject's treatment/study file. Two evaluations are being made in this study. 1. Clinical utility of PEER Interactive where the health outcome of the experimental group will be compared to the outcomes of the control group. 2. Validation of the PEER Interactive outcomes database which is intended to measure post-hoc the health outcomes of participants where the research staff's pharmacotherapy decisions agreed with the output of PEER Interactive.
Who Masked: Participant, Outcomes Assessor
Masking Description: The Subject will be blinded as to study arm assignment and will provide the primary outcome measure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): All subjects will undergo same study procedures. Subjects in the Control Arm will receive treatment as usual by the prescribing clinician/investigator. The prescribing clinician/investigator will not receive the PEER Report of probable medication response for a control arm subject.
- Experimental (Experimental): All subjects will undergo same study procedures. Subjects in the Experimental Arm will receive treatment as usual by the prescribing clinician/investigator. However, the prescribing clinician/investigator will receive the PEER Report of probable medication response for an experimental arm subject. The report will provide additional data/information regarding probable medication response for an experimental arm subject to the prescriber .
  Interventions: Device: The PEER Report

INTERVENTIONS:
Device: The PEER Report — PEER Interactive references a subject's QEEG to a normative and then symptomatic database. By comparing a given subject's QEEG to a database of QEEGs of subjects who have tried and responded to a specific medication, PEER provides useful information regarding the response of neurophysiologically similar subjects to a wide number of medications - providing clinicians with useful information as to medication outcomes before a medication regime is started. Clinicians have also reported that negative findings (in which neurophysiologically similar subjects reported resistant outcomes for certain medications) can be extremely useful in reducing trial and error. It has also been used to help select the medication that best matches the QEEG brainwave pattern.
  Other Names: the PEER Interactive Report; the PEER Online Report
  Arms: Experimental

SUMMARY:
This is a prospective, single-blinded, randomized, multicenter study to evaluate the utility, safety, and efficacy of using PEER Interactive - an EEG-based technology - to inform the prescription of medications to participants with a primary diagnosis of a depressive disorder, with or without comorbidity of non-psychotic behavioral disorders, versus treatment as usual.

DETAILED DESCRIPTION:
This study is observational in nature, in that the participants in the control group will be treated according to treatment as usual and best judgment of the treating clinician. The participants in the experimental group will be treated with adjunctive information provided by the PEER Interactive Report. It is a controlled study in that the schedule of visits, procedures and measurements will be defined by the protocol in order to provide consistent data for both the control and experimental groups.

Participants will be blinded as to presence/use of the PEER Interactive Report and will provide the primary efficacy outcome evaluation. All participants will be randomized into a control or experimental group. All participants will receive a quantitative electroencephalogram (QEEG). For those participants in the experimental group, the research staff will receive an Outcome Report from PEER Interactive. The clinician in the experimental group will use the PEER Interactive Report in the medication prescription process. For the control group, the research staff will not receive an Outcome Report. Outcome Reports for the control group will be sequestered for post-hoc analysis.

The research staff will incorporate the information provided by the Outcome Report from PEER Interactive in their prescription decisions. PEER Interactive provides adjunctive information to assist the treating clinician in the clinical decision process. For the experimental group the research staff is expected to follow the guidance of the subject's PEER Outcome Report as regards to the participant's responsiveness to the on-label medications noted in the Report. Although the study staff is strongly encouraged to use the guidance in the medication decision, prescription of medication is a clinical decision and will be made by the research staff

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 - 65 years of age who speak and read English.
2. Participants able to provide written informed consent to participate in the study.
3. Participants with a primary diagnosis of a DSM-V depressive disorder, including subjects with comorbidity of a non-psychotic behavioral disorder.
4. Participants with comorbidity of mild traumatic brain injury (mTBI) are eligible for inclusion in this study. mTBI will be defined according to best clinical practice guidelines. The subject should have experienced no more than 30 minutes of loss of consciousness, less than a 24 hour alteration in consciousness or mental status, less than 24 hours of post-traumatic amnesia and a Glasgow Coma Scale (best available score in the first 24 hours) of 13 or greater.
5. Participants with comorbidity of post-traumatic stress disorder (PTSD) are eligible for inclusion in this study. A score of 45 or greater on the PTSD Checklist Military/Civilian (PCL-M/C) measurement tool will qualify a subject for inclusion of diagnosis of PTSD as a comorbid condition.
6. Able to stop specified medications, including drugs of abuse, for 5 half-lives of the medication(s). See Appendix B for a list of the five half-life time periods for these medications.

   • The potential subject's primary care physician may be consulted to make these determinations.
7. Able to be washed out of specified medications within 14 days, i.e. 5 half-lives are not longer than 14 days (See Appendix B).
8. Participants will be selected from patients on the psychiatric inpatient ward, partially hospitalized patients, and psychiatric outpatients.
9. Ability to comply with the requirements of the study.

Exclusion Criteria:

1. Male and female subject less than 18 years old or greater than 65 years old
2. Participants who cannot provide written informed consent
3. Diagnosis of a psychotic disorder.
4. History of, or current, open head brain trauma.
5. Subjects with comorbidity of mild traumatic brain injury (mTBI) or traumatic brain injury (TBI) who experienced greater than 30 minutes loss of consciousness, greater than 24 hour alteration in consciousness or mental status, greater than 24 hours of post traumatic amnesia, or a Glasgow Coma Scale (best available score in first 24 hours) of less than 13.
6. Subjects who, in the opinion of the investigator, are unable to washout of specified medications in a period of 14 days or less..
7. History of: craniotomy, cerebral metastases, cerebrovascular accident; current diagnosis of seizure disorder, schizophrenia, schizo-affective disorder, dementia, mental retardation, or major depression with psychotic features; or use of depot neuroleptics in last 12 months.
8. Clinically significant medical illness, including thyroid disorders, which cannot be remediated with medication, e.g. synthroid.
9. Participation in any other therapeutic drug study within 60 days preceding inclusion.
10. Known pregnancy and/or lactation, or intent to become pregnant during this study.
11. Chronic or acute pain requiring prescription pain medication(s) (narcotic or synthetic narcotic).
12. Candidates with any metal, shrapnel or other similar objects in the head that could affect the QEEG.
13. Candidates currently stable and considered to be at Maximum Medical Improvement (MMI) on current medications.
14. Participant has a positive urine drug screen.
15. Participant has active suicidal intent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-06-16 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report 16 Item Questionnaire | Day 0 through study completion, an average of 3 months.
  A proven and accepted survey for measuring symptoms of depression

SECONDARY OUTCOMES:
CHRT-7SR: | Day 0 through study completion, an average of 3 months.
  The Concise Health Risk Tracking Self Report survey (CHRT-7SR) is a 7 question self-report questionnaire that assesses suicidal risk of subjects in clinical practice.
PCL-M/C - if applicable: | Day 0 through study completion, an average of 3 months.
  The PTSD Checklist Military/Civilian is a 17-item self-report measure of the 17 DSM-V symptoms of PTSD. The PCL has a variety of purposes, including: screening individuals for PTSD, diagnosing PTSD, monitoring symptom change during and after treatment. The PCL asks about symptoms in response to "stressful experiences." The Military version is often used with active service members and Veterans. The Civilian version can be helpful when assessing survivors who have symptoms due to multiple events.
Patient-recorded CGI-I (Clinical Global Impressions-Improvement) | Day 0 through study completion, an average of 3 months.
  CGI-I is an assessment by the physician as to the improvement in the subject's mental health. This is a 7-point scale with all subjects beginning with a rating of 4. A ratings of 1 - 3 indicate degrees of improvement, with 1 being 'very much improved, and 3 being 'minimally improved'. A rating of 5 - 7 indicates degrees of worsening, with 5 being 'minimally worse' and 7 being 'very much worse'. A rating of 4 indicates no change from baseline.
Physician-recorded CGI-I (Clinical Global Impressions-Improvement) | Day 0 through study completion, an average of 3 months.
  CGI-I is an assessment by the physician as to the improvement in the subject's mental health. This is a 7-point scale with all subjects beginning with a rating of 4. A ratings of 1 - 3 indicate degrees of improvement, with 1 being 'very much improved, and 3 being 'minimally improved'. A rating of 5 - 7 indicates degrees of worsening, with 5 being 'minimally worse' and 7 being 'very much worse'. A rating of 4 indicates no change from baseline.
CGI-S (Clinical Global Impressions - Severity) - Physician | Day 0 through study completion, an average of 3 months.
  CGI-S is a physician-recorded scale that measures the severity of a subject's mental health. It is a 7-point scale with 1 being 'normal' and 7 being 'extremely mentally ill'.
HAM-D (Hamilton Rating Scale for Depression): | Day 0, Day 15, Day 90
  HAM-D is 17-item interview that will be used as a secondary measure to assess the subject's level of depression

CONTACTS AND LOCATIONS:
Overall Officials: Verner Knott, PhD, Principal Investigator — The Royal, University of Ottawa
Locations (1):
- The Royal Mental Health Center, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Itil TM, Shapiro DM, Herrmann WM, Schulz W, Morgan V. HZI systems for EEG parametrization and classification of psychotropic drugs. Pharmakopsychiatr Neuropsychopharmakol. 1979 Jan;12(1):4-19. doi: 10.1055/s-0028-1094590. PMID 419164
- [Background] Leuchter AF, Cook IA, Marangell LB, Gilmer WS, Burgoyne KS, Howland RH, Trivedi MH, Zisook S, Jain R, McCracken JT, Fava M, Iosifescu D, Greenwald S. Comparative effectiveness of biomarkers and clinical indicators for predicting outcomes of SSRI treatment in Major Depressive Disorder: results of the BRITE-MD study. Psychiatry Res. 2009 Sep 30;169(2):124-31. doi: 10.1016/j.psychres.2009.06.004. Epub 2009 Aug 27. PMID 19712979
- [Result] DeBattista C, Kinrys G, Hoffman D, Goldstein C, Zajecka J, Kocsis J, Teicher M, Potkin S, Preda A, Multani G, Brandt L, Schiller M, Iosifescu D, Fava M. The use of referenced-EEG (rEEG) in assisting medication selection for the treatment of depression. J Psychiatr Res. 2011 Jan;45(1):64-75. doi: 10.1016/j.jpsychires.2010.05.009. Epub 2010 Jul 3. PMID 20598710
- [Result] Iosifescu DV, Greenwald S, Devlin P, Perlis RH, Denninger JW, Alpert JE, Fava M. Pretreatment frontal EEG and changes in suicidal ideation during SSRI treatment in major depressive disorder. Acta Psychiatr Scand. 2008 Apr;117(4):271-6. doi: 10.1111/j.1600-0447.2008.01156.x. Epub 2008 Feb 26. PMID 18307587
- [Result] Knott V, Mahoney C, Kennedy S, Evans K. EEG power, frequency, asymmetry and coherence in male depression. Psychiatry Res. 2001 Apr 10;106(2):123-40. doi: 10.1016/s0925-4927(00)00080-9. PMID 11306251